CLINICAL TRIAL: NCT05218408
Title: A Phase I/IIa Open Label Multicenter, Non-Randomized, Trial to Assess the Safety and Efficacy of CYNK-001in Combination With Recombinant Human Interleukin-2 in Adults With Recurrent Resection Eligible IDH1 Wild-type Glioblastoma
Brief Title: CYNK-001 IV and IC in Combination With IL2 in Surgical Eligible Recurrent GBM With IDH-1 Wild Type
Acronym: CYNK001GBM02
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrolled subjects
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYNK-001-GBM-002
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Astrocytoma, Grade IV; Glioblastoma; Giant Cell Glioblastoma; Glioblastoma Multiforme
Keywords: Interleukin-1; Cyclophosphamide; Fludarabine; immunosuppressive agents; immunological factor; IDH wild type; Surgical GBM; Natural Killer; Cellular Therapy; Allogeneic; Allogeneic stem cell; Ommaya catheter
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: The study will contain two phases for the following objectives •The Phase 1 Dose Escalation will utilize a 3+3 dose escalation design and will evaluate safety, feasibility, and preliminary efficacy of four cohort dose levels of CYNK-001 administered after a 6M IU subcutaneous dose of rhIL-2 for both IV and IC cycles. Up to 21 patients will be enrolled over 4 dosing cohorts in Phase1 and 45 patients enrolled for phase IIa. Cohort 4 will be the safety run for Phase IIa. Cohort 4 in its entirety will be reviewed by the DMC prior to starting Phase 2a portion of this study. Phase 2a will continue to explore efficacy and safety of CYNK-001 in combination with rhIL2 in patients with recurrent resection eligible IDH1 wild-type glioblastoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1Surgical rGBM CYNK-001 infusion ( IV and IC) in combination with IL-2 (Experimental): Phase 1 dose escalation will utilize a 3+3 dose escalation design and will evaluate safety, feasibility, and preliminary efficacy of four cohort dose levels of CYNK-001 administered after a 6M IU subcutaneous dose of rhIL-2 for both IV and IC cycles. Up to 21 patients will be enrolled over 4 dosing cohorts in Phase 1.
  Interventions: Biological: CYNK-001 systemic and Intra cavity administration
- Phase IIa Surgical rGBM CYNK-001 at MPD IV and IC (Experimental): To evaluate efficacy and safety of CYNK-001 administrations in recurrent GBM at maximum tolerated dose for IV and IC per Phase 1 outcome. No patients staggering will be implemented in phase 2a. DMC will review the phase 2a entirely
  Interventions: Biological: CYNK-001 systemic and Intra cavity administration

INTERVENTIONS:
Biological: CYNK-001 systemic and Intra cavity administration — Phase 1 Lymphodepletion Days -5,-4 and -3 Cyclophosphamide 900 mg/m2, Fludarabine 30 mg/m2 and Mesna per SOC
  IL 2 at 6M IU subcutaneous administration:
  For IV cycle ( cycle1) rhIL2 will be administered on Days 1,3,5,8,9,11 and 15 . On days 1, 8 and 15 rhIL-2 will be administered 1 to 3 hours prior to CYNK-001 infusions For IC cycles rhIL2 will be administered 1 to 3 hours prior to each CYNK-001 IC dose.
  CYNK-001 : for IV at 2.4 x10^9 or 3.6 x10^9 cells Days 1,8 and 15
  Tumor resection will take place 7 to 14 day follow by first IC cycle ( Cycle 2) at 100 Million cells or 200 Million cells
  IC cycles 3,4,5 once a week for three weeks , 28 days cycle at100 Million cells or 200 Million cells only for Phase 1 cohort 4 and Phase 2a

SUMMARY:
A Phase 1/2a Open Label Multicenter, Non-Randomized, Trial to Assess the Safety and Efficacy of CYNK-001 in Combination with Recombinant Human Interleukin-2 in Adults with Recurrent Resection Eligible IDH1 wild-type Glioblastoma. For phase I portion, the study objectives to assess the safety and feasibility CYNK-001 in combination with rhIL2 of Intravenous (IV) infusion and Intracavitary (IC) administrations following tumor resection and to establish a maximum tolerated dose (MTD) and a Recommended Phase 2a Dose (RP2D) for IV and IC CYNK-001 administration. For Phase IIa, to evaluate efficacy and safety of CYNK-001 administrations in recurrent GBM as measured by Progression Free Survival at 6 months (PFS6M)

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older of age on the day of signing informed consent.
2. Have had historical or current histologically confirmed isocitrate dehydrogenase 1(IDH1) wild-type glioblastoma and variants as defined by the World Health Organization
3. Patient must have a T1 weighted 3D MRI with Gadolinium enhancement within 14 days prior to lymphodepletion at Day -5
4. Patient must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
5. Radiologically confirmed recurrent glioblastoma at first or second recurrence have contrast enhancing measurable disease with a bidimensional diameter greater than or equal to 10 mm x 10 mm according to RANO and be eligible to undergo tumor resection.
6. Patients must be a candidate to undergo non-emergent surgical resection of the primary target lesion.
7. Multifocal GBM is permissible in the study if there is contiguous T2FLAIR hyperintensity between enhancing lesions on T1 post gadolinium sequences and if in the opinion of the PI surgical resection of the multifocal disease is achievable.

   • NOTE: Multicentric disease with no demonstrated ventricle communication at the time of screening is excluded.
8. The patient must either be on no steroids or on a stable dose of dexamethasone or equivalent no greater than > 2 mg a day for at least 5 days prior to lymphodepletion.
9. Karnofsky performance status (KPS) ≥ 60
10. Have washout periods for prior therapies defined as at five half-lives or (4 weeks) prior to the administration of lymphodepletion whichever is shorter
11. Demonstrate at screening adequate organ function by laboratory values as follows:

    * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
    * Platelet count ≥ 100 x 10^9/L (patient needs to have a minimum of 70 x10^9/L to undergo resection)
    * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2 .5 the upper limit of normal (ULN)
    * Calculated creatinine clearance ≥ 45.0 mL/minute as estimated by Cockcroft-Gault formula
    * Total bilirubin ≤ 1.5 x ULN, unless due to Gilbert's syndrome
    * Total albumin ≥ 3.0 g/dL (30 g/L)
    * Prothrombin Time (PT) ≤1.5 x ULN unless patient is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants
    * activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy if PT or PTT is within therapeutic range of intended use of anticoagulants.
    * Adequate coagulation function defined as INR ≤ 1.5 x ULN, unless the patient is receiving anticoagulant therapy with PT or a PTT/PTT is within therapeutic range.
12. Patients must agree to use a highly effective method of contraception if procreative potential exists from the start of the study until one year after the completion of lymphodepletion for females and 4 months after completion of lymphodepletion for males.

    * A Female of Childbearing Potential (FCBP) is defined as: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

Exclusion Criteria:

1. Midline shift greater than 0.5 cm or pending herniation.
2. Patients who were previously treated with Bevacizumab. The use of Bevacizumab for edema or radiation necrosis treatments may be allowed with prior approval from the medical monitor
3. Anticipated Extent of Resection by volumetric analysis is less than 70%
4. Patients with greater than two recurrences of GBM are excluded
5. Patients with any contraindications to MRIs
6. Treatment with other investigational agents, check point inhibitors and prior immunotherapy such as Vaccine therapy, dendritic cells vaccine within 4 weeks prior to lymphodepletion.
7. Prior radiation therapy within 12 weeks of screening MRI unless there is unequivocal histological confirmation of tumor progression.
8. Patients with known disease in the posterior fossa, gliomatous meningitis, extracranial disease or multicentric enhancing disease. Multicentric disease is defined as discrete sites of contrast enhancing disease without contiguous T2/FLAIR abnormality.

   • NOTE: Satellite lesions that are associated with a contiguous area of T2/FLAIR abnormality as the main lesion(s) may be included.
9. Patients with concurrent use of tumor treating fields (TTF) or laser interstitial thermal therapy (LITT) is excluded. Prior use of TTF or LITT is allowed prior to signing the ICF
10. Patients with current Carmustine wafers. (Patients that agree to remove the Carmustine wafers at the time of tumor resection during the study are allowed in the study)
11. Patents who are receiving systemic steroid therapy > 2 mg of dexamethasone or equivalent total dose per day or any other form of immunosuppressive therapy within 5 days of lymphodepletion.

    • Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients requiring physiological doses of steroids (i.e., adrenal insufficiency or hypopituitarism) not to exceed equivalent of dexamethasone 2 mg will not be excluded from the study.
12. Patients with history of anaphylaxis, angioedema, interstitial pneumonitis, or acute respiratory distress syndrome
13. Active autoimmune disease other than controlled connective tissue disorder or those who are not on active therapy.
14. Any other organ dysfunction (CTCAE Version 5.0 Grade 3 or greater) that will interfere with the administration of the lymphodepletion regimen, rhIL-2, CYNK-001 or the surgical resection as outlined.
15. Known hypersensitivity to cyclophosphamide, fludarabine, Mesna or rhIL-2.
16. Have active or clinically significant cardiac disease including:

    * History or presence of serious uncontrolled cardiac arrhythmias.
    * Clinically significant resting bradycardia.
    * Left ventricular ejection fraction (LVEF) by echocardiogram (ECHO) <50% or multiple gated acquisition scan (MUGA) <45%.
    * Any of the following within 6 months prior to the start of the study treatments: myocardial infarction (MI), severe/unstable angina, congestive heart failure (CHF), transient ischemic attack (TIA).
17. Patients with an SaO2 ≤ 92% on room air.

    • Pulmonary Function Tests may be performed during screening for patients with SaO2 ≤ 92% on room air and based on the clinical judgment of the treating physician, patients with an FEV1 ≥ 50% of predicted and DLCO (corrected) of ≥ 40% of predicted may be enrolled.
18. Has any form of primary immunodeficiency, such as severe combined immunodeficiency disease or acquired immune deficiency syndrome (AIDS).

    • Patients with history of human immunodeficiency virus (HIV) infection must have undetectable HIV ribonucleic acid (RNA).
19. Known active infection with hepatitis B, hepatitis C or other viral infections requiring systemic therapy.
20. Has a QTc prolongation to > 450 millisecond (ms) in males and > 470 ms in females.
21. Is Pregnant or breastfeeding.
22. Received a live vaccine within 30 days prior to lymphodepletion (Day -5).
23. Any other clinically significant medical disease or condition that, in the Principal Investigator's opinion, may interfere with protocol adherence or the patient's ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Phase I-Number of patients experience Dose limiting toxicity (DLT) | 42 days
  Defined as the maximum dose safely administered intravenously or Intracavitary for the treatment of patients with GBM
To establish maximum tolerated dose (MTD) and a Recommended Phase 2a Dose (RP2D) | 42 days
  Defined as the number of patients experience Adverse Events and severity
Phase IIa CYNK-001 efficacy | 6 Months
  To evaluate CYNK-001 efficacy post tumor resection and survival within PFS6 Month

SECONDARY OUTCOMES:
Phase 1-Progression free survival at 6 Months | 6 Months
  is defined as the time from the tumor resection to the date of first documented disease progression determined in accordance with RANO (and iRANO) or death due to any reason, whichever occurs first
Overall survival phase I and IIa | 6,9 and 12 months
  is defined as the time from the tumor resection until the date of death at 6,9 and 12 months

OTHER OUTCOMES:
Progression Free survival Phase I and IIa | 9 and 12 months
  is defined as the time from the tumor resection until the date of death 9 and 12 months (PFS9 and PFS12) post tumor resection
Median Progression Free Survival (mPFS) post tumor resection | 6, 9,12 , 18 and 24 months
  is defined as the median 95% CIs time from the tumor resection until the date of death 9 and 12 months (PFS9 and PFS12) post tumor resection
Median Overall Survival (mOS) post tumor resection | 12 and 24 months
  is defined as the median as the 95%CI time from the tumor resection until the date of death.
Time to Progression (TTP) as measured by RANO | 12 and 24 months
  is defined as the time from the tumor resection to the date of first documented disease progression determined in accordance with RANO(iRANO).
Overall Response Rate (ORR) pre and post tumor resection as measured by RANO | 12 and 24 months
  Defined as the proportion of subjects with best overall response of either complete response (CR) or partial response (PR)
Health Quality of Life assessment using European Organization for Research and Treatment of Cancer-30 with Brain20 module scores | 22, 43, 64,92,120 days
  To assess patient quality of life at baseline and post tumor resection surgery per the schedule of Events using EORTC QLQ C30 and EORTC QLQ BN 20 scale
Evaluation of Neurological Assessment of the Neuro Oncology Scale in Glioblastoma (NANO | 22, 43, 64,92,120 days
  NANO scale provides an objective clinician-reported outcome of neurologic function with high inter-observer agreement
Incidence of Treatment Emergent adverse events (TEAE) | 26 months
  any event not present prior to the initiation of the drug treatment
Incidence and Severity of adverse events (AEs) and clinically significant changes in laboratory values | 26 months
  any untoward or unfavorable medical occurrence in patient during the clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Kilcoyne, MD, Study Director — Celularity inc